CLINICAL TRIAL: NCT00630318
Title: Imaging Protocol Design for Anti-Angiogenesis Tracking With MRI
Brief Title: Testing New Method of Analyzing MR Images
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to accrue enough subjects to analyze data.
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0710-67
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Breast Abnormalities
Keywords: MR scanning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MRI — 15-20 minutes MR imaging

SUMMARY:
Preliminary imaging study to test for future use of this MRI-imaging for evaluating anti-angiogenesis treatment.

DETAILED DESCRIPTION:
The purpose of this study is to develop and evaluate new MR imaging techniques and protocols for non-invasive monitoring of anti-angiogenesis treatment of breast cancer. This feasibility study is a preliminary imaging study to test this imaging protocol on subjects already undergoing MR for clinical purposes.

The specific objective of this research study is to develop and validate both MRI and functional MRI data acquisition methods, task paradigms, and post-processing techniques to ensure reliability of results.

The information derived from this research is intended to be applied to a future study of subjects undergoing experimental anti-angiogenesis drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age 18 years or greater
* Undergoing breast MRI exam

Exclusion Criteria:

* Pregnancy
* Contraindication for MRI on standard screening checklist for clinically indicated examinations (i.e. metal devices/implants; history of claustrophobia)
* History/presence of any of the following to the breast: injury; breast implant; surgical or interventional procedure; clinically significant abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To provide preliminary data for a larger study that this type of imaging can be used to monitor the effectiveness of anti-angiogenic therapy. | After analysis of images

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Clare, MD, Ph.D., Principal Investigator — Indiana University
Locations (1):
- Methodist Hospital, Indianapolis, Indiana, United States